CLINICAL TRIAL: NCT07180121
Title: Information Needs and Supportive Rehabilitation Over Time in Patients Undergoing Cystectomy in Bladder Cancer
Acronym: CaRe
Status: Enrolling by invitation | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Jenny Drott, Associate Professor, Linkoeping University
Other Study IDs: CaRe
Record Dates: First submitted 2025-05-25; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder cancer undergoing radical cystectomy.: Bladder cancer undergoing radical cystectomy.

SUMMARY:
Bladder cancer is one of the diseases that can affect the urinary tract. Globally, it is the tenth most common cancer, with an incidence rate of 9.5 per 100,000 persons per year for men and 2.4 for women. In Sweden, approximately 3,200 patients are diagnosed annually. It predominantly affects the elderly population over 70 years old. Men are more frequently affected, and bladder cancer is now the fourth most common cancer among men in Sweden.

Radical cystectomy is the gold standard treatment for non-metastatic muscle-invasive bladder cancer. The operation involves the removal of the bladder. Most patients are treated with chemotherapy beforehand. A new urinary diversion is created using the small intestine, with the ileal conduit being the most common type. The ureters are connected to the segment of the small intestine, which is then brought out as a stoma on the abdominal wall. Urine will now be collected in a stoma bag. The operation is extensive and can be performed using open or robot-assisted laparoscopic techniques. The average hospital stay for patients undergoing surgery in Sweden is approximately fifteen days.

For patients undergoing cystectomy, their future life is affected by both external and internal physical changes that they need to adapt to. The external physical change with a stoma alters their body appearance, and self-care needs to be performed for the rest of their lives. Self-care, symptoms, and complications can limit patients in their daily lives and negatively impact their social life. The internal physical change affects the internal genital organs and can impact sexual function. This can limit patients' sexual and intimate life.

Receiving a cancer diagnosis is overwhelming. From this moment, a process begins for each individual that involves receiving and absorbing information about the disease and surgery, treatment, and future life. Patients generally have difficulty remembering and absorbing information given during healthcare visits. A cancer diagnosis creates anxiety and is frightening, further impacting what patients remember afterward. Information needs arise when there is a gap between the available information and knowledge compared to what is needed. The patient group feels that their information needs are not met by healthcare personnel during the process from diagnosis to surgery and the immediate time afterward.

Self-care is defined as a process to maintain and uphold health through health-promoting activities and strategies to manage illness. It is a fundamental part of patients' treatment and affects the conditions for adapting to their new everyday life and promotes independent living. Well-functioning self-care contributes to higher health-related quality of life, faster recovery after surgery, reduced risk of complications, less utilization of hospital care leading to reduced healthcare costs, and longer survival. Self-care is an umbrella term that includes self-monitoring and self-management. Self-monitoring involves independently monitoring, interpreting, and assessing whether symptoms require action or contact with healthcare personnel. Self-management is necessary for recovery to manage health problems with troublesome symptoms that arise.

Self-efficacy involves confidence in one's own ability and is significant for adherence to self-care. Empowerment focuses on the ability and responsibility for choices to achieve one's goals and gain control over one's own life. Health literacy is linked to literacy and encompasses a person's knowledge, motivation, and competence to access, understand, assess, and make decisions based on health-related information. Together, these concepts contribute to patients' ability to adapt to their cancer diagnosis and improve their ability to manage treatment-related behavioral changes.

Needs arising from illness and treatment vary over time. They can arise before, during, and sometimes long after the treatment. Continuous, structured mapping of problem areas facilitates the identification of individualized interventions. Cancer rehabilitation promotes health and quality of life and is fundamental to preventing disability, maintaining or regaining previous physical abilities. The level of intervention and education depends on the extent and complexity of the needs and must consider health literacy.

Scientific Purpose of the Project

To explore information needs, health, and supportive rehabilitation in patients with bladder cancer undergoing radical cystectomy.

DETAILED DESCRIPTION:
Specific Objectives

To investigate experiences of information needs in patients with bladder cancer who have undergone cystectomy.

To explore experiences and needs for supportive rehabilitation over time in patients undergoing cystectomy for bladder cancer.

To identify and evaluate patients' information needs, graded health, health literacy, and self-efficacy over time in patients undergoing cystectomy for bladder cancer.

ELIGIBILITY:
Inclusion criteria:

- Patients >18 years who have undergone cystectomy at two hospitals and are Swedish-speaking.

Exclusion criteria:

- Patients with cognitive impairment or cognitive memory loss will be screened using the 4AT.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years who have undergone cystectomy at two hospitals and are Swedish-speaking.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Information needs | 1 year
  EORTC QLQ-INFO25

OTHER OUTCOMES:
Questionnarie to assess symptoms and health | 1 year
  longitudinal measurements of symptoms and health, questionnarie in line with "my care plan cancer"
health litteracy | baseliine
  Validated instrument; s-fhl and s-chl
Self efficacy | baseline
  The General Self-Efficacy Scale (GSE)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Linköping, Sweden